CLINICAL TRIAL: NCT02746939
Title: Student Behavior Outcomes in Fitness and Nutrition Integrated Science Education Outreach (InSciEd Out, ISEO)
Brief Title: Student Outcomes in Fitness and Nutrition ISEO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing change
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher Pierret, Assistant Professor - Department of Biochemistry and Molecular Biology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-001162
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: program evaluation; health literacy; fitness; nutrition; education
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-curriculum assessment (No Intervention): Assessments will be administered to 3rd and 4th grade students prior to receiving curriculum training in fitness and nutrition.
- Post-curriculum assessment (Experimental): Assessments will be administered to 3rd and 4th grade students (matched from pre-curriculum assessment) after receiving 4-6 week InSciEd Out Fitness and Nutrition Curriculum.
  Interventions: Behavioral: InSciEd Out Fitness and Nutrition Curriculum

INTERVENTIONS:
Behavioral: InSciEd Out Fitness and Nutrition Curriculum — Science curriculum is designed in partnership with 3rd and 4th grade teachers and InSciEd Out scientists. The curriculum is designed to focus on inquiry driven science, and also aims to decrease high risk behaviors that can lead to obesity in the students.
  Arms: Post-curriculum assessment

SUMMARY:
The study is designed to examine whether curriculum, designed in partnership with teachers at Moreland Elementary school in West St. Paul and Mayo Clinic InSciEd Out scientists, is able to influence the behavior and health literacy of students. This information will be collected in surveys before and after the students are given the curriculum during the school day.

DETAILED DESCRIPTION:
The research will implement a short battery of two survey inventories to measure student outcomes under InSciEd Out Fitness and Nutrition curriculum that is currently administered in 3rd and 4th grade at Lincoln K-8 Choice School. One is a grade-level adapted version of the National Youth Physical Activity and Nutrition Survey (NYPANS) authored by the United States Center for Disease Control (CDC). The other is a grade-level adapted version of the Newest Vital Sign (NVS) health literacy assessment authored by Pfizer and adapted by Dr. Linda Aldoory at the University of Maryland.

These assessments will help inform the health promotion activities of the InSciEd Out partnership within Lincoln K-8 Choice in Rochester, Minnesota (MN) and Moreland Elementary in West St. Paul, MN who originally wrote the curriculum. These assessments will be key to curricular revision and expansion to other schools that partner with InSciEd Out. As such, this study is a single cohort, internally controlled pre-post assessment of an existing behavioral intervention. Pending pilot study success, future follow-up studies are projected to be parallel-group, nonrandomized clinical trials of a treatment school versus a control school with grade levels expansion. This study will inform activities within the InSciEd Out network inside Rochester Public Schools (RPS), where grades Kindergarten through 2nd and 5th through 8th curricula is currently being built. Previously RPS-approved Mayo Clinic Institutional Review Board (IRB) #13-003263 describes the format of InSciEd Out programming in detail, but the general framework of this study operates upon an established partnership between InSciEd Out researchers and Lincoln K-8 Choice/Moreland Elementary administrators, teachers, students, and parents.

IRB#13-003263 describes the format of InSciEd Out programming in detail, but the general framework of this study operates upon an established partnership between InSciEd Out researchers and administration, teachers, and students at Lincoln K-8 Choice Elementary.

ELIGIBILITY:
Inclusion Criteria:

* Students attending 3rd and 4th grade classes at Lincoln K-8 Choice Elementary School in Rochester, MN or Moreland Elementary School in West St. Paul, MN who assent to the study

Exclusion Criteria:

* Students attending 3rd and 4th grade classes at Lincoln K-8 Choice Elementary School in Rochester, MN or Moreland Elementary School in West St. Paul, MN whose parents chose to opt-out of the study or who do not assent to the study

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with completion of ISEO Fitness and Nutrition Curriculum | 9 months
  students will undergo 4-6 weeks of ISEO fitness and nutrition curriculum as part of their 3rd or 4th grade coursework. Classroom teachers will decide when to administer the curriculum, but should be completed by January 2017 in our target classrooms.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Pierret, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No